CLINICAL TRIAL: NCT05883111
Title: HPV Methylation Self-testing Pilot in Transgender Individuals
Brief Title: HPV Self-testing in Transgender Individuals
Acronym: Self-TI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 319364
Record Dates: First submitted 2023-04-24; First posted 2023-05-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HPV Infection
Keywords: Transgender; Trans men; Trans women; Non-binary individuals
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans men and non-binary people with a cervix (Other): Participants will have a clinician-collected cervical screening sample and then collect the following self-samples for research: Vaginal swab, Anal swab, Oral rinse, and Urine sample for the detection of HPV detection.
  Interventions: Diagnostic Test: HPV DNA methylation assay
- Trans women and non-binary people (Experimental): Participants will collect the following self-samples for research in the clinic: Vaginal swab, Anal swab, Oral rinse, and Urine sample for the detection of HPV detection. Participants will collect the following self-samples for research at home: Vaginal swab, Anal swab, and Oral rinse sample for the detection of HPV detection.
  Interventions: Diagnostic Test: HPV DNA methylation assay

INTERVENTIONS:
Diagnostic Test: HPV DNA methylation assay — HPV DNA methylation assay to detect HPV positivity, HPV genotype, and HPV methylation.

SUMMARY:
Human papillomavirus (HPV) is a common virus that spreads through skin-to-skin contact. Some HPV types can cause changes in cells that lead to cancer and are known as 'high-risk' HPV (hrHPV). hrHPV is linked to cancers of the cervix (opening of the womb), throat, and anus (exit of the bowel).

It is not known if transgender people (individuals whose gender identity does not align with their sex assigned at birth) are at increased risk of hrHPV or cancers caused by hrHPV compared to cisgender people (individuals whose gender identity does align with their birth sex). There is also little knowledge about HPV in the vagina for transgender women who have surgery to make one.

Transgender men may be at higher risk of cervical cancer than cisgender women because they are less likely to go for screening. This can be because of physical discomfort and emotional distress during screening when a swab is taken directly from the cervix.

The investigators seek to examine how common hrHPV is in transgender people in different parts of the body. In the study, participants will take swabs from the vagina and anus, a urine sample, and use mouthwash. Transgender men will also have an extra swab taken by a clinician as part of routine cervical screening. This is to see if the swab from the vagina is as good as the one from the cervix for finding cells that might lead to cancer. Participants will also take an online survey to measure the acceptability of self-sampling compared to clinician sampling.

This research can inform HPV prevalence and decision-making about HPV screening among transgender people.

ELIGIBILITY:
Inclusion criteria for trans men and non-binary adults with a cervix:

* Identify as transgender or non-binary
* Be between 25 - 65 years of age
* Be registered with a general practitioner
* Have an intact cervix
* Have used testosterone therapy within the last year
* Be willing, and able to understand and consent to study procedures

Inclusion Criteria for trans women and non-binary adults :

* Identify as transgender or non-binary
* Be 18 years of age or older
* Have undergone vaginoplasty by any method at least 1 year ago
* Be willing, and able to understand and consent to study procedures

Exclusion Criteria:

* Have a variation of sex characteristics (also known as a disorder of sex development)
* Have an allergy to any of the ingredients in the oral rinse (Scope)
* Be diagnosed with, or under investigation for, an inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease). This does not include irritable bowel syndrome - participants with this are eligible to enroll.
* Be a member of a vulnerable population, which includes pregnant people, fetuses, children, prisoners, or anyone unable to independently offer consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender and gender diverse identities.
Enrollment: 100 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of self-sampling in clinic | Baseline
  Feasibility of self-sampling in clinic as measured by the proportion of completed and returned self-samples.
Acceptability of self-sampling in clinic | Baseline
  Acceptability of self-sampling in clinic as indicated by high satisfaction on an online survey
Feasibility of self-sampling at home | 1 month follow-up
  Feasibility of self-sampling at home as measured by the proportion of completed and returned self-samples.
Acceptability of self-sampling at home | 1 month follow up
  Acceptability of self-sampling at home as indicated by high satisfaction on an online survey

SECONDARY OUTCOMES:
HPV concordance between vaginal self-sample and clinician-collected cervical swab | Baseline
  Concordance HPV positivity, overall and by genotype, from self-collected vaginal samples to clinician-collected cervical samples in trans men and nonbinary adults with a cervix.
HPV correlation between self-samples taken at clinic and in home among trans women and non-binary people. | Baseline and 1 month follow up
  HPV correlation between self-samples taken at clinic and in-home among trans women and non-binary people.

OTHER OUTCOMES:
HPV correlation between self-samples at each site | Baseline and 1 month follow up
  HPV correlation between self-samples at each site (vaginal, anal, oral, and urine) in each arm.
Performance of HPV methylation assay | Baseline
  Comparison of the performance of HPV methylation testing from self-collected samples to clinician-collected samples for the detection of cervical precancer in trans men and non-binary adults with a cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Jackson, PhD, Principal Investigator — National Cancer Institute (NCI); Alison M Berner, MBBS, PhD, Principal Investigator — Queen Mary University of London
Locations (3):
- United Kingdom (3):
  - University Hospitals Sussex NHS Foundation Trust Sexual Health Service, Brighton
  - Ambrose King Centre, Barts Health NHS Trust, London
  - CliniQ, Caldicott Centre, Kings College Hospitals, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson SS, O'Callaghan S, Ward E, Orkin CM, Clarke MA, Berner AM. Rationale and design of the Self-TI Study protocol: a cross-sectional human papillomavirus self-testing pilot study among transgender adults in England. BMJ Open. 2024 Jul 4;14(7):e086099. doi: 10.1136/bmjopen-2024-086099. PMID 38964803